CLINICAL TRIAL: NCT02948595
Title: Video Feedback Versus Verbal Feedback in Simulated Laparoscopic Vaginal Cuff Closure
Brief Title: Video Feedback Versus Verbal Feedback
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Principal Investigator, Naomi Y Swanson, Assistant Professor, Department of Obstetrics and Gynecology, University of New Mexico
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 16-096
Record Dates: First submitted 2016-07-21; First posted 2016-10-28 (Estimated); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Resident Surgical Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Video feedback then verbal feedback (Experimental): Video feedback followed by structured verbal feedback
  Interventions: Other: Video feedback followed by structured verbal feedback
- Verbal feedback then video feedback (Experimental): Structured verbal feedback followed by video feedback
  Interventions: Other: Structured verbal feedback followed by video feedback

INTERVENTIONS:
Other: Video feedback followed by structured verbal feedback — Video feedback followed by structured verbal feedback
  Arms: Video feedback then verbal feedback
Other: Structured verbal feedback followed by video feedback — Structured verbal feedback followed by video feedback
  Arms: Verbal feedback then video feedback

SUMMARY:
The long term goal of our research is to develop a curriculum for Obstetrics and Gynecology resident physicians that regularly employs use of video assessment to improve surgical skills. Regular use of video feedback may enable improved self-assessment and allow for formal documentation of proficiency. The overall objective is to compare the use of video feedback to use of structured verbal feedback in the simulated task of laparoscopic vaginal cuff closure.

ELIGIBILITY:
Inclusion Criteria:

* Resident Physician in the Department of Obstetrics and Gynecology

Exclusion Criteria:

* Not a resident physician in the Department of Obstetrics and Gynecology

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2016-11-18 (Actual); Primary Completion 2017-05-03 (Actual); Study Completion 2017-05-03 (Actual)

PRIMARY OUTCOMES:
Improvement in ob/gyn resident physician self-efficacy as measured by self-efficacy questionnaire in video versus verbal feedback for simulated laparoscopic vaginal cuff closure | up to 18 months
  Resident physicians will report their self-efficacy in completion of simulated laparoscopic vaginal cuff closure using an adaptation of a previously validated self-efficacy questionnaire. Their self-efficacy will be compared after completion of the task incorporating verbal feedback from a proctor to completion of the task incorporating review of video feedback provided by proctor.

SECONDARY OUTCOMES:
Improvement in time of simulated laparoscopic vaginal cuff closure with video versus verbal feedback | up to 18 months
  Resident physicians will be timed (in minutes) for completion of simulated laparoscopic vaginal cuff closure. Time will be compared in completion of the task after verbal feedback from a proctor versus completion of task after video feedback from a proctor.
Improvement in skill of simulated laparoscopic vaginal cuff closure as measured by Objective Structured Assessment of Technical Skills (OSATS) global rating scale with video versus verbal feedback | up to 18 months
  Two advanced gynecologic laparoscopists will review the films of the tasks for each resident physician. They will rate level of skill for each participant based on Objective Structured Assessment of Technical Skills (OSATS) global rating scale. The reviews will generate two scores for each participant: the score for the task completed after the resident receives verbal feedback and the score for the task completed after the resident receives video feedback. The two scores will then be compared for each participant.

IPD SHARING:
Plan to Share IPD: No